CLINICAL TRIAL: NCT06818487
Title: Ganyan-1 in Dry Eye: A Randomized Clinical Trial
Brief Title: Ganyan-1 in Dry Eye
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DED_TCM_2024
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye; TCM
Keywords: Dry eye; TCM; RCT
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ganyan1 (Experimental)
  Interventions: Drug: Ganyan1; Drug: Sodium Hyaluronate
- 1/2Ganyan1 (Experimental)
  Interventions: Drug: Sodium Hyaluronate; Drug: 1/2Ganyan1
- Placebo (Placebo Comparator)
  Interventions: Drug: Sodium Hyaluronate; Drug: Placebo

INTERVENTIONS:
Drug: Ganyan1 — During the treatment period, participants will receive the following Chinese herbal granules, including Chrysanthemum, Dendrobium, Salvia miltiorrhiza, Gypsum Fibrosum, and Goji berries, administered twice daily at a dose of 10 g per time for a duration of 4 weeks.
  Arms: Ganyan1
Drug: Sodium Hyaluronate — Participants received 0.1% sodium hyaluronate eye drop
Drug: 1/2Ganyan1 — During the treatment period, participants will receive the following Chinese herbal granules, including Chrysanthemum, Dendrobium, Salvia miltiorrhiza, Gypsum Fibrosum, and Goji berries, administered twice daily at a dose of 5 g per time for a duration of 4 weeks.
  Arms: 1/2Ganyan1
Drug: Placebo — Participants will receive the following placebo Chinese herbal granules, administered twice daily at a dose of 10 g per time for a duration of 4 weeks.
  Arms: Placebo

SUMMARY:
Ganyan -1 for the patients with dry eye

DETAILED DESCRIPTION:
Objective: Ganyan-1 for the patients with dry eye Methods: The investigators enrolled 219 patients at Beijing Tongren Hospital. Patients completed questionnaires at baseline, week2, week4, week8, week12, and week16.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 and Age <=70, complaint of DED symptoms for 6 months or longer at screening.

3. ocular surface disease index (OSDI) score of 25 or higher. 4. tear film breakup time (TFBUT) of 5 seconds or less. 5. Schirmer I test without anesthesia of 5 mm or more at 5 minutes. 6. CFS score of 4 or higher.

Exclusion Criteria:

1. History systemic autoimmune diseases and ocular/periocular malignancy.
2. Clinically relevant slitlamp findings or abnormal lid anatomy.
3. Active ocular allergies and active infection.
4. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
OSDI | Baseline, week 2, 4, 8, 12 and 16
  The Ocular Surface Disease Index (OSDI) includes 12 questions grouped by poor symptoms and visual disturbance (light sensitivity, eyes feel gritty, painful or sore eyes, blurred vision or poor vision); visual function/tasks (problems when reading, driving at night, working on a computer or watching TV); and environmental questions (problems in windy conditions, places/ areas with low humidity or areas that are air conditioned). The scores range from 0 to 100. On the basis of the score, the patient's symptoms can be categorized as normal (0-12), mild dry eye (13-22), moderate dry eye (23-32), or severe dry eve (33-100).

SECONDARY OUTCOMES:
TBUT | Baseline, week 2, 4, 8, 12 and 16
  Tear breakup time (TBUT) is a clinical test used to assess for evaporative dry eye disease. To measure TBUT, fluorescein is instilled into the patient's tear film and the patient is asked not to blink while the tear film is observed under a broad beam of cobalt blue illumination. The TBUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film, as seen in this progression of these slit lamps' photos over time. A TBUT under 10 seconds is considered abnormal.
Schirmer | Baseline, week 2, 4, 8, 12 and 16
  The Schirmer test is objectively used to measure tear secretion without anesthetized. A healthy eye should wet more than 10 mm of the standard filter strip in 5 minutes. The travel rate along the test strip is proportional to the tear production rate.
SF-36 | Baseline, week 2, 4, 8, 12 and 16
  36-Item Short Form Health Survey (SF36) measures quality of life on the basis of eight dimensions or concepts that are frequently used in health studies. These eight dimensions are estimated from eight subscales that examine physical functioning (SF36-PF), role functioning-physical (SF36-RP), bodily pain (SF36-BP), general health (SF36- GH), vitality (SF36-VT), social functioning (SF36-SF), role functioning-emotional (SF36-RE), mental health (SF36-MH) and reported health transition (SF36-HT). Item responses were ranaina from 0 (best) to 100 (worst), with hiaher scores are equivalent to areater severity of better quality of life.
SAS | Baseline, week 2, 4, 8, 12 and 16
  The SAS is a 20-item self-report instrument designed to assess anxiety symptoms in clinical and research settings. This scale ranges from 20 to 80, with lower scores indicating better self-reported mental health and fewer anxiety symptoms.
SDS | Baseline, week 2, 4, 8, 12 and 16
  Medical Outcomes from study 20-Item Self-Rating Depression Scale. This scale range is 0-100 with lower scores indicating better self-reported mental health.
OQAS II | Baseline, week 2, 4, 8, 12 and 16
  Medical Outcomes from the OQAS II Visual Quality Assessment The OQAS II measures visual quality using several optical parameters. Scores are generated based on metrics like the Modulation Transfer Function (MTF) and Objective Scatter Index (OSI). The scale ranges from 0-100, with lower scores indicating better optical quality and fewer distortions. Change is calculated as the score at follow-up time points (e.g., post-treatment or surgery) minus the baseline score.